CLINICAL TRIAL: NCT02560298
Title: InterAACT - An International Multicentre Open Label Randomised Phase II Advanced Anal Cancer Trial Comparing Cisplatin Plus 5-Fluorouracil Versus Carboplatin Plus Weekly Paclitaxel in Patients With Inoperable Locally Recurrent or Metastatic Disease
Brief Title: Cisplatin and Fluorouracil Compared With Carboplatin and Paclitaxel in Treating Patients With Inoperable Locally Recurrent or Metastatic Anal Cancer
Acronym: InterAACT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA2133; NCI-2015-00771 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA2133; 13/LO/1463; CCR 3847; 2013-001949-13; InterAACT CCR 3847; 3847; EA2133 (Other: ECOG-ACRIN Cancer Research Group); EA2133 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Anal Basaloid Carcinoma; Anal Canal Cloacogenic Carcinoma; Anal Squamous Cell Carcinoma; Metastatic Anal Canal Carcinoma; Recurrent Anal Canal Carcinoma; Stage IIIB Anal Canal Cancer; Stage IV Anal Canal Cancer
MeSH Terms: conditions — Anal Canal Carcinoma; Anus Neoplasms | interventions — Capecitabine; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Fluorouracil; dehydroftorafur; Paclitaxel; Taxes

ARMS (2):
- Arm A (cisplatin, fluorouracil or capecitabine) (Experimental): Patients receive cisplatin IV over 1-4 hours on day 1 and fluorouracil IV continuously over 24 hours on days 1-4. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity. Patients with complications associated with the central venous access which prevent further infusion of fluorouracil and only after discussion with the Chief Investigator receive capecitabine BID on days 1-4.
  Interventions: Drug: Capecitabine; Drug: Cisplatin; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment
- Arm B (paclitaxel, carboplatin) (Experimental): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Capecitabine
  Other Names: Ro 09-1978/000; Xeloda
  Arms: Arm A (cisplatin, fluorouracil or capecitabine)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm B (paclitaxel, carboplatin)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm A (cisplatin, fluorouracil or capecitabine)
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Arm A (cisplatin, fluorouracil or capecitabine)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm B (paclitaxel, carboplatin)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase II trial studies how well cisplatin and fluorouracil work compared with carboplatin and paclitaxel in treating patients with anal cancer that cannot be removed by surgery, has come back at or near the same place as the primary tumor, or spread to other places in the body. Drugs used in chemotherapy, such as cisplatin, fluorouracil, carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether cisplatin and fluorouracil are more effective than carboplatin and paclitaxel in treating anal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate best overall response rate (ORR).

SECONDARY OBJECTIVES:

I. Overall survival (OS). II. Progression free survival (PFS). III. Disease control rate (DCR) (stable disease [SD] or better) at 12 and 24 weeks.

IV. Best ORR of non-irradiated lesions. V. Anti-tumor activity and magnitude of response as captured by waterfall plot analyses.

VI. Toxicity. VII. Quality of life (QOL). VIII. Feasibility of conducting a multicenter international study on squamous cell carcinoma of the anus (SCCA) and recruit within a reasonable time frame.

TERTIARY OBJECTIVES:

I. Explorative biomarker analysis.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive cisplatin intravenously (IV) over 1-4 hours on day 1 and fluorouracil IV continuously over 24 hours on days 1-4. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity. Patients with complications associated with the central venous access which prevent further infusion of fluorouracil and only after discussion with the Chief Investigator may receive capecitabine twice daily (BID) on days 1-4.

ARM B: Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable, locally recurrent or metastatic disease (tumor resectability should be assessed by a local surgeon or multidisciplinary team)
* Histological or cytological confirmation of epidermoid anal carcinoma (includes squamous, basaloid and cloacogenic lesions) from the primary tumor or a newly diagnosed recurrent/metastatic lesion
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1
* Previous definitive chemo-radiation is permitted for early stage tumors (cisplatin-based chemotherapy [chemo]-radiation is permitted but only if tumor progression/relapse occurs after 6 months from treatment completion)
* Previous systemic chemotherapy is permitted if administered as induction treatment (=< 2 cycles) before definitive chemoradiotherapy for early stage disease and there is no evidence of tumor progression during or after treatment completion
* Human immunodeficiency virus positive (HIV+) patients will be considered eligible if they are on highly active anti-retroviral therapy (HAART) and have a cluster of differentiation (CD)4 count of >= 200/ul (HIV+ patients who are on HAART and have a CD4 count < 200/ul are eligible if the plasma viral load is below the level of detection according to the local assay)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/l
* Platelets >= 100 x 10^9/l
* Hemoglobin (Hb) >= 9 g/dl for males and >= 8 g/dl for females
* Creatinine clearance >= 50 ml/minute
* Serum bilirubin =< 1.5 x upper limit of normal (ULN)
* Alanine transaminase (ALT) or aspartate transaminase (AST) =< 3 x ULN (if liver metastases are present, serum transaminases =< 5 x ULN are permitted)
* Fertile men and women must agree to take adequate contraceptive precautions during, and for at least six months after therapy
* Life expectancy of at least 3 months

Exclusion Criteria:

* Tumors of adenocarcinoma, melanoma, small cell and basal cell histology are excluded
* Locally recurrent tumor which is amenable to curative resection (as deemed by a local surgeon or multidisciplinary team)
* Tumor relapse/progression within 6 months of completion of a cisplatin-based chemoradiotherapy regimen for the treatment of early stage tumors
* Previous administration of > 2 cycles of systemic chemotherapy as induction treatment before definitive chemoradiotherapy for early stage disease
* Tumor progression during or immediately after completion of =< 2 cycles of systemic chemotherapy as induction treatment before definitive chemoradiotherapy for early stage disease
* Previous use of systemic chemotherapy or other investigational drugs for the treatment of inoperable locally recurrent or metastatic tumors (previous use of radiotherapy in this setting is not an exclusion criterion if: 1) non-irradiated target tumor lesions are present at randomization for the purpose of tumor response assessment or 2) in the absence of non-irradiated target tumor lesions, progression of the irradiated tumor lesions according to the RECIST criteria version 1.1 is documented)
* Current or recent (within 30 days of first study dosing) treatment with another investigational drug or participation in another investigational study
* Documented or symptomatic brain metastases and/or central nervous system metastases or leptomeningeal disease
* Major surgery performed < 28 days from treatment start
* Palliative radiotherapy completed =< 7 days from treatment start
* Clinically significant (i.e. active) cardiac disease (e.g. symptomatic coronary artery disease, uncontrolled cardiac arrhythmia, or myocardial infarction within the last 6 months); any history of clinically significant cardiac failure
* History of interstitial lung disease (e.g. pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest computed tomography (CT) scan
* HIV+ patients who are not on HAART or have a CD4 count of < 200/ul in the presence of detectable plasma viral load according to the local assay
* Known history of active hepatitis B or hepatitis C infection
* Serious active infection requiring intravenous (i.v.) antibiotics at enrollment
* Other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer
* Other clinically significant disease or co-morbidity that may adversely affect the safe delivery of treatment within this trial
* Known hypersensitivity to any of the study drugs or excipients
* Known peripheral neuropathy > grade 1 (absence of deep tendon reflexes as the sole neurological abnormality does not render the patient ineligible)
* Pre-existing hearing impairment
* Patients planning for a live vaccine
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Best ORR defined as the percentage of patients achieving confirmed partial (PR) or complete responses (CR) as per RECIST v1.1 | Up to 3 years
  The ORR will be summarized as the percentage (including 95% confidence intervals) of responders and presented by treatment group and will be compared (as exploratory endpoint) between treatment groups using a chi-squared test.

SECONDARY OUTCOMES:
Anti-tumor activity and magnitude of response | Up to 3 years
  Anti-tumor activity and magnitude of response will be captured by waterfall plot analyses. The percentage change in tumor size from baseline to the time of best response will be plotted by patients (ordered from worst to best) and bars colored according to best response.
Best ORR of non-irradiated lesions defined as the percentage of patients achieving confirmed PR or CR as per RECIST v1.1 of non-irradiated sites of disease | Up to 3 years
  The ORR of non-irradiated lesions will be summarized as the percentage (including 95% confidence intervals) of responders and presented by treatment group and will be compared (as exploratory endpoint) between treatment groups using a chi-squared test.
Changes in QOL | Baseline to up to 3 years
  QOL will be evaluated using the European Organization for Research and Treatment of Cancer Core Quality of Life and EuroQOL-5 dimension-5 level questionnaires. Differences from baseline will be compared between arms of the study using the two sample t-test or Wilcoxon non-parametric method as appropriate.
DCR defined as CR, PR, or SD assessed according to RECIST criteria v1.1 | At 24 weeks post treatment start
  DCR will be summarized as the percentage (including 95% confidence intervals) of responders and presented by treatment group and will be compared (as exploratory endpoint) between treatment groups using a chi-squared test.
DCR defined as CR, PR, or stable disease (SD) assessed according to RECIST criteria v1.1 | At 12 weeks post treatment start
  DCR will be summarized as the percentage (including 95% confidence intervals) of responders and presented by treatment group and will be compared (as exploratory endpoint) between treatment groups using a chi-squared test.
Feasibility in terms of proportion of centers that successfully recruit at least one patient | Up to 36 months
  The proportion of centers engaging will be presented with 95% confidence intervals.
Feasibility in terms of recruitment rate | Up to 36 months
  The recruitment rate will be calculated overall centers and by country and center.
OS | From the date of randomization to the date of death from any cause, assessed up to 12 months
  The Kaplan Meier estimates of OS over time and median OS with associated 95% confidence intervals will be presented by treatment and (as exploratory endpoint) compared using a log rank test. Cox multivariate regression analysis will be used (as exploratory analysis) to calculate the hazard ratio between treatments along with its 95% confidence interval. The treatment effect will be adjusted for the stratification factors and other identified prognostic factors (e.g. time to disease relapse & whether pre-treated with platinum) in a multivariate setting.
PFS | From the date of randomization to the date of confirmed clinical/radiological progression or death from any cause, assessed up to 12 months
  The Kaplan Meier estimates of PFS over time and median PFS with associated 95% confidence intervals will be presented by treatment and (as exploratory endpoint) compared using a log rank test. Cox multivariate regression analysis will be used (as exploratory analysis) to calculate the hazard ratio between treatments along with its 95% confidence interval. The treatment effect will be adjusted for the stratification factors and other identified prognostic factors (e.g. time to disease relapse & whether pre-treated with platinum) in a multivariate setting.
Proportion of patients experiencing grade 3-5 toxicity graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 3 years
  The proportion of patients experiencing grade 3-5 toxicity will be compared on a regimen basis using the chi-squared test. Fisher's exact test will be used when expected cell frequencies are < 5.
Sensitivity analysis of ORR | Up to 3 years

OTHER OUTCOMES:
Changes in expression of tumor biomarkers | Up to 3 years
  Multivariate analyses will be performed to evaluate the effect of known prognostic factors and biomarkers on outcomes observed.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Eng, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States